CLINICAL TRIAL: NCT02718131
Title: A Study of INFUSE Bone Graft (Recombinant Human Bone Morphogenetic Protein-2/Absorbable Collagen Sponge) in the Treatment of Tibial Pseudarthrosis in Neurofibromatosis 1 (NF1)
Brief Title: A Study of INFUSE Bone Graft (BMP-2) in the Treatment of Tibial Pseudarthrosis in Neurofibromatosis Type 1 (NF1)
Acronym: NF107-BMP2
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient enrollment to meet the statistical requirements
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: The Children's Tumor Foundation (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, Bruce Korf, MD, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NF107; W81XWH-12-1-0155 (Other Grant/Funding Number: Department of Defense, US Army); G140004 (Other: FDA IDE); 507821 (Other: Medtronic)
Record Dates: First submitted 2016-03-07; First posted 2016-03-24 (Estimated); Results first posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-09

CONDITIONS: NF1; Congenital Pseudarthrosis of Tibia
Keywords: Tibial Pseudarthrosis
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- INFUSE Bone Graft (BMP-2) (Active Comparator): Children with NF1 and tibial pseudarthrosis who require surgery will have the INFUSE bone graft added to their surgical protocol. After a standard surgical approach of resection of abnormal pseudarthrotic tissue, placement of a rigid intramedullary rod (of the surgeon's choice) and placement of autogenous bone graft from the iliac crest; in addition, the INFUSE bone graft in the form of a collagen sponge will be wrapped around the tibia during the surgical process.
  Interventions: Device: INFUSE Bone Graft (BMP-2)
- Control Group (Placebo Comparator): Children with NF1 and tibial pseudarthrosis who require surgery will receive the standard surgical protocol only. This includes resection of abnormal pseudarthrotic tissue, placement of a rigid intramedullary rod (of the surgeon's choice) and placement of autogenous bone graft from the iliac crest.
  Interventions: Procedure: Control Group

INTERVENTIONS:
Device: INFUSE Bone Graft (BMP-2) — The INFUSE bone graft, containing BMP-2 on a collagen sponge, will be wrapped around the tibia during the surgical process.
  Arms: INFUSE Bone Graft (BMP-2)
Procedure: Control Group — The control group will receive the standard surgical protocol, without addition of the INFUSE device.
  Arms: Control Group

SUMMARY:
The current study proposes adding BMP-2 (INFUSE), an anabolic agent, at the surgical site of TPA (tibial pseudarthrosis) repair in children with NF1, compared to a control group of patients treated surgically without BMP-2. The following Specific Aims will be addressed: 1) to determine if use of an osteogenic agent (BMP-2) at the time of surgical repair of TPA in NF1 patients will result in improved bone healing; 2) to document safety of BMP-2 in a pediatric NF1 population; and 3) to collect, process, and preserve biologic specimens at the time of surgery for future studies.

DETAILED DESCRIPTION:
A randomized study will be performed by a multi-center group of the NF Consortium. A total of 54 patients will be randomized for treatment with or without INFUSE Bone Graft at the time of surgical repair. For all patients, a standard surgical procedure will be used, including: resection of pseudarthrosis tissue; placement of a rigid intramedullary rod; and placement of autogenous bone graft from iliac crest. For patients in the BMP group, the INFUSE device containing BMP-2 will in addition be applied intraoperatively to the osteotomy site. Fracture union will be determined by scoring of radiographs (RUST score) for cortical bone fusion and callus formation at the osteotomy site. RUST score at 12 months post-surgery will be the primary outcome measure to determine efficacy. Secondary measures will include determination of time to healing (months); quality of life measures; functional walking measures; and incidence of refracture after surgery. This study, once successfully completed, will determine if use of INFUSE Bone Graft improves healing of tibial pseudarthrosis in NF1 and will document safety issues. Regardless of results, the better performing of the two groups (control or BMP) will be able to serve as a much-needed control arm for future studies of additional targeted therapeutic agents for NF1-related bone disease. An international working group of orthopaedic surgeons and NF specialists has been formed and is committed to successful completion of this trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NF1 using the NIH Consensus Conference criteria. In addition to tibial pseudarthrosis, one or more of the following diagnostic criteria for NF1 must be present:
* Six or more cafe'-au-lait spots (≥ 0.5cm prepubertal; ≥ 1.5cm postpubertal)
* Freckling in the axilla or groin Optic pathway glioma
* Two or more iris Lisch nodules
* Two or more neurofibromas or one plexiform neurofibroma
* A first-degree relative with NF1
* Patients must have tibial pseudarthrosis that has the potential to cause significant morbidity. Radiographic findings (AP & lateral leg radiographs) must support the diagnosis of tibial pseudarthrosis with chronic non-union.
* Age between 2 years and 18 years of age at time of study entry.
* Performance Level: Karnofsky ≥ 50 percent for patients > 10 years of age and Lansky ≥ 50 percent for patients or ≤ 10 years of age.

Prior Therapy:

* Patients who have undergone 1 previous surgery for tibial pseudarthrosis repair will be eligible to enter the study if they have refracture.
* Use of BMP-2 in the prior surgery is permitted, however patients with prior exposure must be screened for antibodies to BMP-2, bovine collagen, and rhBMP-2 neutralizing antibodies.
* Prior use of BMP-2 is allowed but will be recorded as a possible compounding factor.
* Patients who have had 2 or more prior surgeries for pseudarthrosis repair are ineligible

Absence of Tumors:

* Patients must undergo thorough physical examination of the leg undergoing surgery. If physical exam is equivocal for presence of tumors, then a normal MRI of the lower extremity will be required before eligibility is met.
* If there is evidence of plexiform neurofibroma or nodular neurofibroma of > 3 cm diameter on the ipsilateral leg, then they are ineligible for the study.
* Organ Function Requirements
* Adequate bone marrow function defined as:

  * Absolute neutrophil count (ANC) > 1500/
  * µl Platelet count > 100,000/
  * µl Hemoglobin ≥ 10.0 gm/dL

Adequate renal function defined as:

* maximum serum creatinine of 1.5 mg/dL OR
* a creatinine clearance≥70ml/min/1.73m2.

Adequate renal function defined as:

* maximum serum creatinine of 1.5 mg/dL OR
* a creatinine clearance ≥ 70ml/min/1.73m2.

Adequate liver function defined as:

* Total bilirubin < 1.5 X upper limit of normal for age, and SGPT (serum glutamic pyruvic transaminase, ALT) < 2 X upper limit of normal for age
* Serum Vitamin D level ≥ 10 ng/ml

Exclusion Criteria:

* Lack of documentation for a diagnosis of NF1
* Tibial fracture without evidence of pseudarthrosis or tibial dysplasia
* Tibial dysplasia/bowing without fracture or pseudarthrosis
* Plexiform neurofibroma of any size, or nodular neurofibroma of > 3 cm diameter involving the ipsilateral leg, including the hip
* If presence of plexiform is suspected but not certain on physical exam, MRI of the leg may be indicated to rule this out.
* History of MPNST (malignant peripheral nerve sheath tumor) or any malignancy other than asymptomatic and stable optic nerve glioma
* Optic nerve glioma that has resulted in precocious puberty or visual impairment of any degree
* Visual impairment from any cause
* Precocious puberty from any cause
* Hypertension other than mild essential hypertension controlled with medication
* Metastatic disease of any kind
* Inadequate neurovascular status in the involved limb that may jeopardize healing
* Active or known prior infection at the pseudarthrosis site
* Active systemic infection
* Other injury or condition that prevents ambulation or completion of study assessments
* Two or more prior surgeries for tibial pseudarthrosis
* Bilateral tibial dysplasia
* Selection of a surgical approach that does not include prescribed surgical intervention, which must include removal of pseudarthrosis tissue, placement of an intramedullary rod using the Williams approach, and autogenous bone graft from the iliac crest distributed at the osteotomy site
* Normal ipsilateral fibula without planned fibular osteotomy at time of surgery
* Allergy to bone morphogenetic protein
* Allergy to bovine collagen products
* Positive antibody titers to BMP-2, bovine collagen, or BMP-2 neutralizing antibodies prior to surgery
* History of using any of the following medications, regardless of dose, for at least 1 month, within 3 months of enrollment: Anabolic agents, Glucocorticoids (does not include inhaled glucocorticoids), Growth hormone, Parathyroid hormone (PTH)
* Need for postoperative medications that could interfere with bone healing of the implant, such as steroids, (but not including low-dose aspirin or routine perioperative anti-inflammatory drugs)
* Untreated endocrine abnormality, such as hypothyroidism, parathyroid hormone disorder
* Severe Vitamin D deficiency with serum 25-OH (hydroxy) Vitamin D < 10 ng/ml (25 nmol/l) Patients with Vitamin D levels < 10 ng/ml may be treated with Vitamin D and reconsidered for enrollment when levels are sufficient
* Females who are sexually active without use of effective contraception
* Females who are pregnant or breastfeeding

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce R. Korf, MD, PhD, Study Chair — Univ. of Alabama at Birmingham
Locations (16):
- United States (15):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Lurie Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana Unversity, Indianapolis, Indiana
  - Johns Hopkins, Baltimore, Maryland
  - Children' Hospital Boston and Massachusetts General Hospital, Boston, Massachusetts
  - Children' Hospital Boston, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - New York University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Scottish Rite Hospital for Children, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
- The Children's Hospital at Westmead, Westmead, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- INFUSE Bone Graft (BMP-2): Standard surgery plus BMP-2
- Control Group: Standard surgery without BMP-2
Period: Overall Study
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group
Started | 5 | 0
Completed 12 Months | 2 | 0
Completed | 2 | 0
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Data was incomplete. Patient was inevaluable | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomization resulted in 0 participants for the Control Group
Groups:
- Total: Total of all reporting groups
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 0 | 5
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.4 (3.1) |  | 3.4 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 2 |  | 2
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 |  | 4
RUST score [Median (Full Range); unit: scores on a scale] — The RUST scale (Radiographic Union Score for Tibial fractures; RUST) is a measure of tibial fracture healing. Score is based on radiographic evaluation of the bone cortex based on AP and lateral xrays. Four cortices of tibial bone are each given a score of 1 to 3, with 1=no healing, 2=some callus present, and 3=healing of the bone cortex. The 4 scores are totaled for a total score range of 4 to 12. For this study, a total RUST score of 9 to 12, with at least 2 evaluable cortices having a score of 3, is considered to be healed. Scores of 5 to 8 = partial healing, and a score of 4 = no healing.
  scores on a scale | 11 [10 to 12] |  | 11 [10 to 12]

OUTCOME MEASURES:

1. Primary Outcome: RUST Score
Description: The RUST scale (Radiographic Union Score for Tibial fractures; RUST) was developed in 2010 as a measure of tibial fracture healing and has been validated in the NF1 population. This was used as the primary outcome measure in this trial. The score is based on radiographic evaluation of the bone cortex based on AP (anterior-posterior) and lateral xrays. Four cortices of tibial bone seen in these views are each given a score of 1 to 3, with 1 representing no healing, 2 representing some callus present, and 3 representing healing of the bone cortex. The 4 scores are totaled, to give a total score range of 4 to 12. For the purpose of this study, a total RUST score of 9 to 12, with at least 2 evaluable cortices having a score of 3, is considered to be healed. Scores of 5 to 8 are considered to represent partial healing, and a score of 4 is considered to be no healing.
Time Frame: 12 mos post surgery. The score at 12 mos post surgery will be used to determine success of healing and is the score reported.
Population: The population consisted of 2 evaluable participants. Three (3) participants withdrew for various reasons (see participant flow). The study was closed for further enrollment due to poor recruitment. The study was closed after the last participant completed study procedures.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group
Number analyzed (Participants) | 2 | 0
score on a scale | 12 [12 to 12] |

2. Secondary Outcome: Average Time to Healing in Months
Description: Time to healing is determined by RUST scores calculated at 3 month intervals after surgery. The first time point at which a score of 9 to 12 is achieved on the RUST Scale will be considered the time to complete healing. One time point is reported which is the time point of first healing.
Time Frame: Baseline through 12 months post-surgery.
Population: as for outcome 1
Measure: Median (Full Range); unit: months
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group
Number analyzed (Participants) | 2 | 0
months | 4.5 [3 to 6] |

3. Secondary Outcome: Refracture Rate
Description: Numbers of patients with refracture within 1 year after surgery.
Time Frame: 12 months post-surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group
Number analyzed (Participants) | 2 | 0
Participants | 0 | 0

4. Secondary Outcome: Long-term Refracture
Description: Numbers of patients with refracture over long-term follow up of up to 10 years.
Time Frame: annually, up to 10 years post-surgery
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group
Number analyzed (Participants) | 1 | 0
Participants | 0 | 0

5. Secondary Outcome: Ten Meter Timed Walk
Description: Time (seconds) to perform the Ten Meter Timed Walk. Assessed at 6 and 12 months after surgery. Both 6 month and 12 month reported.
Time Frame: Assessed at 6 and 12 months after surgery. Month 12 reported.
Population: as for outcome 1
Measure: Median (Full Range); unit: seconds
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group
Number analyzed (Participants) | 2 | 0
seconds
  6 month measure | 20.2 [7 to 33.3] |
  12 month measure: number analyzed (Participants) | 1 | 0
  12 month measure | 11.3 [11.3 to 11.3] |

6. Secondary Outcome: Pain Intensity
Description: Pain Intensity was measured using the Faces Pain Scale-Revised (FPS-R) for patients aged 4 years and older. This is a self-report pain scale, where children chose one of 6 faces to indicate their current pain. Scores range from 0 to 10, with 0 representing no pain (happy face) and 10 representing the most pain.
Time Frame: measured at post-op visits at 6 weeks, 3 mos, 6 mos, and 12 mos after surgery
Population: Participants were all too young to report on this scale (younger than age 4 years). No results are reported.
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Quality of Life Score - The Upper Extremity and Physical Function Core Scale
Description: Quality of Life (QOL) was measured during the study using the Pediatric Outcome Data Collection Instrument (PODCI), a validated scale developed by the American Academy of Orthopaedic Surgeons to measure outcomes in orthopedic interventions. The Parent-report form, which was used for this study, consists of 86 Likert-format questions, covering 5 domains (Upper extremity and physical function; transfer and basic mobility; sports/physical functioning; pain/comfort; and happiness scales). In addition, a Global Functioning Scale is computed. Scores for each subscale range from 0 to 100, with lower scores representing better quality of life.
Time Frame: Assessed at 6 and 12 months after surgery. Month 12 reported.
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group
Number analyzed (Participants) | 2 | 0
score on a scale | 76 [40 to 100] |

8. Secondary Outcome: Quality of Life Score - The Transfer and Basic Mobility Core Scale
Description: as for outcome 7
Time Frame: Assessed at 6 and 12 months after surgery. Month 12 reported.
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group
Number analyzed (Participants) | 2 | 0
score on a scale | 61 [43 to 85] |

9. Secondary Outcome: Quality of Life Score - The Sports and Physical Functioning Core Scale
Description: as for outcome 7
Time Frame: Assessed at 6 and 12 months after surgery. Month 12 reported.
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group
Number analyzed (Participants) | 2 | 0
score on a scale | 65 [11 to 81] |

10. Secondary Outcome: Quality of Life Score - The Pain/Comfort Core Scale
Description: as for outcome 7
Time Frame: Assessed at 6 and 12 months after surgery. Month 12 reported.
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group
Number analyzed (Participants) | 2 | 0
score on a scale | 75 [22 to 100] |

11. Secondary Outcome: Quality of Life Score - The Happiness Core Scale
Description: as for outcome 7
Time Frame: Assessed at 6 and 12 months after surgery. Month 12 reported.
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group
Number analyzed (Participants) | 2 | 0
score on a scale | 90 [80 to 100] |

12. Secondary Outcome: Quality of Life Score - The Global Functioning Scale
Description: as for outcome 7
Time Frame: Assessed at 6 and 12 months after surgery. Month 12 reported.
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group
Number analyzed (Participants) | 2 | 0
score on a scale | 65 [44 to 91] |

ADVERSE EVENTS:
Time Frame: 1 year after surgery
Description: The population consisted of 2 evaluable participants. Three (3) participants withdrew for various reasons (see participant flow). The study was closed for further enrollment due to poor recruitment. The study was closed after the last participant completed study procedures. No participants were randomized to the control group.
Arm/Group | INFUSE Bone Graft (BMP-2) | Control Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/5 | 0/0
Other Adverse Events (participants affected / at risk) | 2/5 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INFUSE Bone Graft (BMP-2) (N=5) | Control Group (N=0)
Surgical and Medical procedure - revision of Rush rod (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INFUSE Bone Graft (BMP-2) (N=5) | Control Group (N=0)
New fracture tibia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
In June 2019 at the recommendation of the study protocol chairs, the study was closed for enrollment with plans to terminate the study after the last patient completed study procedures. Therefore limited data is available for analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT02718131/Prot_SAP_000.pdf